CLINICAL TRIAL: NCT04597645
Title: Effects of Therapeutic Elastic Band Training on Body Composition and Physical Capacity in Adults With Prader-Willi Syndrome
Brief Title: Prader-Willi Syndrome Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCRD-TPE-109-55
Record Dates: First submitted 2020-08-21; First posted 2020-10-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-02

CONDITIONS: Prader Labhart Willi Syndrome; Body Weight Changes; Sarcopenia
Keywords: Prader Willi Syndrome; Body composition; Sarcopenia; Resistance training; Physical capacity
MeSH Terms: conditions — Prader-Willi Syndrome; Body Weight Changes; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic band (EB) (Experimental): EB group participants who are attending sheltered employment will received Elastic Thera band training program two times per week (once supervised and guided by a trained physical therapist and the other supervised by educational trainer) over 16 weeks for a total of 32 sessions.
  Interventions: Other: Therapeutic elastic band resistance training
- Control group (CG) (No Intervention): Control group participants will receive usual care.

INTERVENTIONS:
Other: Therapeutic elastic band resistance training — A16-week therapeutic program using Elastic Thera Band will be taught. The exercises are designed to train specific major muscle groups, strengthen the motivation of participants, and facilitate home-based compliance. The program will be performed two times per week (once supervised and guided by a trained physical therapist and the other supervised by educational trainers) over 16 weeks for a total of 32 sessions. Each session supervised by a physical therapist last for 60 minutes, including a 5-minute warm-up consisting of light-intensity aerobic and dynamic stretching exercises, followed by 50 minutes of EB exercise and a 5-minute period of cool-down and static stretching exercises.
  Arms: Elastic band (EB)

SUMMARY:
Adults aged over 18 years, with the diagnosis of Prader-willi syndrome will be recruited through the hospital's outpatient clinic for either as intervention group receiving therapeutic elastic band training, or as control group receiving usual care for a total of 16 weeks. Body composition, physical capacity, and serum changes will be assessed before and after the intervention.

DETAILED DESCRIPTION:
Participants that fulfill the inclusion criteria will be assigned into one of the two arms: elastic band intervention group (EB) or control group (CG). Both groups will received a baseline: dual X-ray absorptiometry body composition, physical capacity, and serum markers examinations. EB will then receive a 16-week progressive elastic band resistance exercise training, while the CG will receive usual care. After the 16 weeks from the baseline assessment, a followed-up: dual X-ray absorptiometry body composition, physical capacity, and serum examinations will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old.
* Genetically diagnosis of Prader-willi syndrome.
* Must be able to follow and understand mandarin instructions and cooperate to the exercise assessments and/or training.

Exclusion Criteria:

* Prader-willi syndrome individuals unable to sit, stand and walk independently which make physical capacity assessment difficult.
* Severe arthritis, fracture, or other musculoskeletal deformities that interfere with exercise training.
* Severe cognitive impairment who cannot read, write the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in lean tissue mass and adipose tissue mass | Baseline and 4 month follow up
  Lean tissue mass and adipose tissue mass will be determined by dual energy x-ray absorptiometry (DXA) (Hologic Densitometer Discovery A, USA).
Change in body mass index | Baseline and 4 month follow up
  Body mass index will be calculated as the body mass in kilograms divided by the square of the height in meters.

SECONDARY OUTCOMES:
Change in grip muscle strength | Baseline and 4 month follow up
  A baseline hydraulic dynamometer will be used to assess the grip muscle strength. The upper extremity muscle quality (ratio of muscular strength to muscle mass) will be calculated by dividing handgrip strength by arm lean mass.
Change in 30-second sit to stand test | Baseline and 4 month follow up
  The 30-second sit to stand test assesses endurance by counting the number of sit to stand ups achieved.
Change in timed up and go test | Baseline and 4 month follow up
  The timed up and go test measures the time required to rise from a chair, walk a 3-meter-long line on the floor, turn around, walk back, and sit down again.
Change in two minute step up test | Baseline and 4 month follow up
  The two minute step up test measures aerobic endurance by having the subject marching in place for two minutes, lifting alternatively the knees to a midway between patella and iliac crest height of a tape (marked at the wall).
Change in Berg balance scale | Baseline and 4 month follow up
  Berg balance scale assesses simple mobility function tasks (sit unsupported, sit-to-stand, stand to sit, stand unsupported, transfer, stand with eyes closed and feet together) and more difficult balance tasks (turn to look behind, retrieve object from floor, turn 360 degrees, reach forward with an outstretched arm, tandem stand, place alternate foot on stool, and single leg stand). It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4. A maximum scoring of 56 indicates functional balanced, while scoring< 45 indicates higher risk of falling.
Change in lipid profile | Baseline and 4 month follow up
  Measurements of serum levels of total cholesterol, triglyceride, low-density lipoprotein, and high-density lipoprotein will be determined using biochemical automatic analyzer according to the manufacturer's recommendations and established methods in the literature.
Change in fasting glucose | Baseline and 4 month follow up
  Measurements of serum levels of fasting glucose will be determined using biochemical automatic analyzer according to the manufacturer's recommendations and established methods in the literature.
Change in glycated hemoglobin | Baseline and 4 month follow up
  Measurements of the glycated hemoglobin (HbA1c) of fasting glucose will be determined using biochemical automatic analyzer according to the manufacturer's recommendations and established methods in the literature.

OTHER OUTCOMES:
Change in appendicular skeletal muscle mass and lower extremity skeletal muscle mass | Baseline and 4 month follow up
  The appendicular skeletal muscle mass (ASM) will be obtained from the dual energy x-ray absorptiometry (DXA) (Hologic Densitometer Discovery A, USA) measurement, excluding the bone mass from the mass of the extremities, from which fat mass is already excluded. ASM (kg)=lean body mass of extremity - bone mass of extremity.
  The lower extremity skeletal muscle mass (LESM) will be obtained from the dual energy x-ray absorptiometry (DXA) (Hologic Densitometer Discovery A, USA) measurement, by excluding the bone mass of the lower extremity, from which fat mass is already excluded. LESM (kg)=lean body mass of lower extremity - bone mass of lower extremity.
Change in skeletal muscle mass index and lower extremity skeletal muscle mass index | Baseline and 4 month follow up
  Skeletal muscle mass index (SMI) (%) will be calculated using the values measured via the dual energy x-ray absorptiometry (DXA) (Hologic Densitometer Discovery A, USA) as follow= ASM (kg)/body weight (kg)×100 Lower extremity skeletal muscle mass (LESM) (%) will be calculated using the values measured via the dual energy x-ray absorptiometry (DXA) (Hologic Densitometer Discovery A, USA) as follow= LESM (kg)/lower extremity body weight (kg)×100)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Chiu, MD, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) is not planned to be shared.